CLINICAL TRIAL: NCT06965699
Title: Testing the Effect of a Plant-based, Protein-dense Sauce (ProSauce) on Metabolic Availability of Essential Amino Acids and Gut Fullness and Satiety in Older Adults
Brief Title: The Effect of a Plant-based, Protein-dense Sauce on Essential Amino Acid Concentrations and Gut Fullness in Older Adults
Acronym: ProSauce
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: ProSauce Uo
Record Dates: First submitted 2025-04-23; First posted 2025-05-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Malnutrition Elderly; Protein Malnutrition
Keywords: plant-based protein sauce; older adults; amino acid metabolic availability; appetite regulation
MeSH Terms: conditions — Kwashiorkor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProSauce (Experimental)
  Interventions: Dietary Supplement: ProSauce
- standard sauce (Placebo Comparator)
  Interventions: Dietary Supplement: low-protein sauce

INTERVENTIONS:
Dietary Supplement: ProSauce — 10g additional protein from ProSauce
  Arms: ProSauce
Dietary Supplement: low-protein sauce — Commercially available standard low-protein sauce
  Arms: standard sauce

SUMMARY:
The goal of this clinical trial is to determine whether meals fortified with plant-based high protein sauce (ProSauce) provide better metabolic availability of essential amino acids compared to meals with standard lower-protein sauce without resulting in excessive gut fullness and satiety. The main questions it aims to answer are:

Does meals with high-protein sauce deliver better metabolic availability of amino acid profile? Does this high-protein sauce also not lead to excessive appetite suppression due to its liquid form? Researchers will compare high protein sauce to a commercially available standard low protein sauce.

Participants will consume two meals, either protein-fortified or standard low-protein sauce, in a randomised order with at least a one-week washout period between each meal. The investigators will collect venous blood samples over a 6-hour postprandial period to measure plasma essential (and non-essential) amino acid and insulin concentrations. The investigators will also measure appetite-related hormones from venous plasma and assess subjective appetite using a visual analogue scale, taken in parallel with the blood sample time points.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 and over
* Living independently in the community
* Capacity to provide informed consent
* Non-smoking (vaping is considered smoking)
* No known medical conditions that might influence the study outcomes, e.g., heart disease, diabetes mellitus, obesity, disthyroidism and other endocrinopathies and renal failure
* Not taking any medications that might influence the study outcomes e.g., taking anabolic steroids or corticosteroids long term
* No clinically diagnosed eating disorders
* No severe dislike or allergy to any of the study food
* No hospitalisations in the last 6 months
* Not dieting and weight stable for 3 months before the study (< 3 kg change in weight)

Exclusion Criteria:

* Age < 60y
* Smoking
* Food allergies
* Cognitive and mobility issues
* Hospitalisation in the last 6 months
* Known medical conditions that might influence the study outcomes
* Taking medications that influence the study outcomes

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Concentrations of essential amino acids | Essential amino acid concentrations at time points of baseline, immediately after breakfast (t =0 minute) and t = 20, 40, 60, 90, 120, 180, 240, 300, 360 minutes.
  Baseline and postprandial plasma amino acid concentrations will be measured to provides valuable insights into protein digestion and absorption.

SECONDARY OUTCOMES:
Concentrations of appetite-related gut hormones | Appetite-related gut hormones will be measured at time points of baseline, immediately after breakfast (t =0 minute) and t = 20, 40, 60, 90, 120, 150, 180, 210, 240 minutes.
  Plasma appetite-related hormones i.e., acylated ghrelin, PYY, GLP-1, CCK, will be measured at certain time points via cannulation.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Bowtell, Prof, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No